CLINICAL TRIAL: NCT01295606
Title: Cefazolin Pharmacokinetics: Elimination Clearance in Neonates
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S52907; 2010-024319-15 (EudraCT Number)
Record Dates: First submitted 2010-12-07; First posted 2011-02-14 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2010-12

CONDITIONS: Prophylaxis
Keywords: cefazolin; prophylaxis; pharmacokinetics; newborn
MeSH Terms: interventions — Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cefazolin, antibiotic prophylaxis (No Intervention): All included patients will received iv cefazolin
  Interventions: Drug: Cefazolin

INTERVENTIONS:
Drug: Cefazolin — iv cefazolin (50mg/kg, 3 times a day) will be given as a routine prophylaxis treatment
  Other Names: Kefzol

SUMMARY:
To document cefazolin disposition (concentration/time profile, protein binding, metabolism, renal elimination characteristics) and its covariates in neonates following intravenous administration of the drug at induction of anesthesia, prior to an invasive procedure

To evaluate if optimalisation of cefazolin dose regimen during neonatal life is needed

DETAILED DESCRIPTION:
Prospective, single-center, open label study on the pharmacokinetics of iv cefazolin administration in neonates admitted in the neonatal intensive care unit, University Hospitals Leuven, Belgium.

Patients will be included after signed informed consent of the parents.

Our aim is to include 40 neonates. Cefazolin has been selected for this study as it is routinely administered in neonates undergoing invasive procedures in our unit. At this stage, we only have the intention to document pharmacokinetics and covariates based on the current clinical practice and therefore will not interfere with either clinical indication, or with dosing as prescribed by the attending physician.

Drug administration and collection of samples will be obtained to the current clinical and nursing standard procedures.

Routine clinical care for scheduled invasive procedures in neonates in our unit is intravenous administration of cefazolin as follows:

* 50 mg/kg, 3 times a day
* an extra dose of 50mg/kg is given after 3 hours for operations longer than 3 h
* each time one dose/day is excluded for neonates with body weight <2000 g and postnatal age (PNA) <7 days,
* for invasive operations (e.g. open-heart surgery, laparotomy) the prophylactic administration of cefazolin may be continued for 3-5 days following the completion of surgery.

The antibiotic agent should be administered 30 minutes to 1 hour prior to the start of surgery so that adequate antibiotic levels. Cefazolin is administered to the neonate, through a peripherally inserted venous catheter, during 30 minutes.

Blood will be collected in heparinised tubes through an indwelling arterial line, or deep venous access, always when other routine blood samples are collected for clinical purposes (pO2, pCO2, pH).

Urine samples will be collected through a bladder catheter in patients in whom a bladder catheter is available for clinical indications.

Pharmacokinetic analysis A population pharmacokinetics approach will be used, hereby comparing the data on PK already reported in adults or older children and the newly collected data during neonatal life.

ELIGIBILITY:
Inclusion Criteria:

* signed parental informed written consent
* neonates to whom cefazolin is administered by intravenous route for clinical indications (invasive procedure)

Exclusion Criteria:

* known cefazolin intolerance

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of iv cefazolin in neonates | up to 24 h following the first dose administration (in surgical procedures with forein-body implantation up to 48 h following the first dose administration)

SECONDARY OUTCOMES:
Optimalisation of cefazolin dose regimen during neonatal life | up to 24 h following the first dose administration (in surgical procedures with forein-body implantation up to 48 h following the first dose administration)

CONTACTS AND LOCATIONS:
Overall Officials: Karel Allegaert, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven

REFERENCES:
- [Derived] Elkayal O, Allegaert K, Spriet I, Smits A, Seghaye MC, Charlier C, Dreesen E. Population pharmacokinetics of cefazolin in maternal and umbilical cord plasma, and simulated exposure in term neonates. J Antimicrob Chemother. 2021 Nov 12;76(12):3229-3236. doi: 10.1093/jac/dkab329. PMID 34499720